CLINICAL TRIAL: NCT02911298
Title: An Open Label, Single-site Pharmaco-Scintigraphic Phase I - Study in Healthy Subjects to Evaluate the Gastrointestinal Transit and Release Profile of Radio-labelled Metronidazole Benzoate Capsules
Brief Title: Pharmaco-Scintigraphic Study to Evaluate the Release Profile of Metronidazole Benzoate Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tillotts Pharma AG (Industry)
Collaborators: Swiss Commission for Technology and Innovation (Other); University of Basel (Other); University Hospital, Basel, Switzerland (Other); SocraTec R&D GmbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TP-CTI-01
Record Dates: First submitted 2016-09-02; First posted 2016-09-22 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mucoadhesive formulation (Experimental): A single dose of 100 mg Metronidazole Benzoate gastro-resistant capsule with radio-labelled mucoadhesive formulation is administered to subject in fasted state
  Interventions: Drug: Metronidazole Benzoate gastro-resistant capsule with radio-labelled mucoadhesive formulation
- Non-mucoadhesive formulation (Active Comparator): A single dose of 100 mg Metronidazole Benzoate gastro-resistant capsule with radio-labelled non-mucoadhesive formulation is administered to subject in fasted state
  Interventions: Drug: Metronidazole Benzoate gastro-resistant capsule with radio-labelled non-mucoadhesive formulation

INTERVENTIONS:
Drug: Metronidazole Benzoate gastro-resistant capsule with radio-labelled mucoadhesive formulation
  Arms: Mucoadhesive formulation
Drug: Metronidazole Benzoate gastro-resistant capsule with radio-labelled non-mucoadhesive formulation
  Arms: Non-mucoadhesive formulation

SUMMARY:
This is a Phase I, open label, single-site trial to evaluate the in vivo release characteristics in the gastrointestinal tract of metronidazole benzoate capsules designed to disintegrate in the large intestine. This will be examined by means of metronidazole plasma levels and scintigraphic images in healthy subjects. Overall, nine subjects will be evaluated for each formulation prototype. Two formulation prototypes will be investigated. Each subject will receive one radio-labelled capsule only.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects, male or non-pregnant, non-lactating females, between 18 and 55 years old. Females of child bearing potential must have a negative urine pregnancy test prior to the intake of study drug, and must use a hormonal (oral, implantable or injectable) or a double barrier method of birth control throughout the study. Females unable to bear children must have documentation of such in the source records (i.e., tubal ligation, hysterectomy, or post-menopausal with as a minimum of one year since the last menstrual period).
2. Ability of subject to participate fully in all aspects of this clinical trial.
3. Voluntary signed informed consent must be obtained and documented.
4. Accept not to use any kind of tobacco, including cigarettes nor E-Cigarettes or pipe smoking, nicotine replacements nor oral tobacco and not to consume any alcohol or drugs during screening, treatment and following two days.

Exclusion Criteria:

1. Participating in a clinical study involving investigational drugs or dosage forms within the previous 30 days.
2. Radiation exposure from clinical trials, including that from the present study and from diagnostic X-ray but excluding background radiation, exceeds 5 mSv in the last five years. No subject whose occupational exposure is monitored will participate in the study.
3. Any nuclear medicine procedure prior to study day 1 that might interfere with the scintigraphic images that are acquired.
4. Clinically significant deviation of biochemistry or haematology parameters from the normal range
5. History of gastrointestinal surgery, with the exception of appendectomy unless it was performed within the previous 12 months.
6. Clinically relevant cardiovascular, renal, hepatic, metabolic, autoimmune, pulmonary and particularly gastrointestinal diseases, especially peptic ulceration, gastrointestinal bleeding, ulcerative colitis, Crohn's disease or Irritable Bowel Syndrome (within the previous 12 months).
7. Acute diarrhoea or constipation in the 14 days before the predicted first study day. If screening occurs >14 days before first study day, this criterion is to be determined on the first study day. Diarrhoea will be defined as the passage of liquid faeces and/or a stool frequency of greater than three times per day. Constipation will be defined as a failure to defecate more frequently than every three days.
8. History of adverse reaction or allergy to metronidazole or any study drug or formulation components/ingredients.
9. Hypersensitivity to imidazole derivatives
10. History of any malignancy removed or adequately treated.
11. History of alcohol or drug abuse.
12. Donation of blood (or plasma) within the previous three months and donation of Plasma the last 14 days.
13. Over-the-counter (OTC) and prescription medication (including laxatives, vitamins and natural herbal remedies including St. John's Wort) between screening visit (visit 1) and completion of the study. Occasional paracetamol or acetyl-salicylic acid is permitted.
14. Ingestion of grapefruit juice, coffee, caffeine containing beverages on treatment day.
15. Failure to satisfy the Investigator to participate for any other reason.
16. Known allergy to crustaceans (due to Chitosan)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-11-25 (Actual); Primary Completion 2017-03-06 (Actual); Study Completion 2017-03-06 (Actual)

PRIMARY OUTCOMES:
Scintigraphic analysis of time of capsule disintegration | 3 days
Scintigraphic analysis of location of capsule disintegration | 3 days
Transit time of the released granules after capsule disintegration | 3 days

SECONDARY OUTCOMES:
Maximal plasma concentration (Cmax) | 3 days
Time to reach Cmax (Tmax) | 3 days
Area under the concentration-time curve | 3 days
Elimination rate constant (k) | 3 days
Apparent terminal half-live (t½) | 3 days
Lag time (t-lag) | 3 days
Time of first measurable concentration after dosing | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Haschke, MD, Principal Investigator — University Hospital Basel, Phase I Research Unit
Locations (1):
- University Hospital Basel, Phase I Research Unit, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No